CLINICAL TRIAL: NCT02193191
Title: Safety and Efficacy Trial of Escalation of Plerixafor for Mobilization of CD34+ Hematopoietic Progenitor Cells and Evaluation of Globin Gene Transfer in Patients With Sickle Cell Disease
Brief Title: Escalation of Plerixafor for Mobilization of CD34+ Hematopoietic Progenitor Cells and Evaluation of Globin Gene Transfer in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sanofi (Industry); New York Blood Center (Other); Weill Medical College of Cornell University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-229
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease
Keywords: Plerixafor; 13-229
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor

ARMS (1):
- Plerixafor (Experimental): Patients will receive a single dose of subcutaneous plerixafor with peripheral blood studies at approximately 0-2 hours before, approximately 6-12 hours after, and approximately 20-48 hours after plerixafor administration, with leukapheresis in the last 3 patients on the protocol. Collected HPCs will be transferred to the MSKCC CTCEF to determine if the HPCs are amenable to transduction with a lentiviral vector encoding the normal ß- globin gene.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor

SUMMARY:
The purpose of this research study is to test the safety and efficacy of a drug called Plerixafor. Plerixafor is approved by the US FDA for use in increasing blood stem cell counts before collection in cancer patients. It is not yet approved for patients with sickle cell disease. The investigators want to find out if Plerixafor can be used to increase cell counts in patients with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed and measurable Sickle Cell Disease, defined by SS or Sβ thalassemia confirmed by hemoglobin fractionation.
* ≥ 18 to 65 years of age
* Patient must have a ECOG performance status ≤2 or Karnofsky score > 70%
* Patients must have acceptable organ and marrow function as defined below:

  * WBC ≥ 3,000/μL
  * ANC ≥ 1,500/μL
  * platelets ≥150,000//μL
  * Hemoglobin ≥ 6 gm/dL
  * Calculated creatinine clearance ≥ 60ml/min * *Using the Cockcroft-gault equation [140 - Age(yrs)] [Weight(kg)] x 0.85 if Female 72 [Serum Creatinine (mg/dL]
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Patients who are:

  * Receiving or received treatment with an investigational agent within 4 weeks prior to entering the study OR
  * have not recovered from adverse events due to agents administered more than 4 weeks earlier as determined by the treating physician.
* Patients with ALT(SGPT) > 2.5 X upper limit of normal
* Patients with a creatinine clearance of < 60 ml/min
* Patients who have uncontrolled illness including, but not limited to:

  * Ongoing or active infection
  * Emergency room admission or hospitalization in the past 14 days
  * Major surgery in the past 30 days
  * Medical/psychiatric illness/social situations that would limit compliance with study requirements as determined by the treating physician.
* Female patients who are pregnant or breast-feeding
* Patients with active hepatitis B, hepatitis C, or HIV infection
* Patients with poor cardiac function as defined by an ejection fraction < 40% are excluded due to potential poor tolerance of the fluid shifts with leukapheresis (only for patients enrolled on second phase of protocol for Leukapheresis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
safety | up to 30 days
  Safety is assessed using a dose limiting toxicity (DLT) endpoint. Definition of a DLT is the occurrence of any of the below events that meets the following criteria: The occurrence of a vasoocclusive crisis requiring hospitalization, acute chest syndrome, CNS acute event, or any other disease related ischemic-based adverse event (AE) should be considered as a DLT, if occurring in the 48 hours DLT observation period.
efficacy | ≥ 30/ul at either 6-12 hours or 24-48 hours post plerixafor.
  Efficacy is defined as 100% of evaluable patients reaching a PB CD34 concentration ≥ 30/uL.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tamari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York

REFERENCES:
- [Derived] Boulad F, Zhang J, Yazdanbakhsh K, Sadelain M, Shi PA. Evidence for continued dose escalation of plerixafor for hematopoietic progenitor cell collections in sickle cell disease. Blood Cells Mol Dis. 2021 Sep;90:102588. doi: 10.1016/j.bcmd.2021.102588. Epub 2021 Jun 15. PMID 34166998
- [Derived] Avecilla ST, Boulad F, Yazdanbakhsh K, Sadelain M, Shi PA. Process and procedural adjustments to improve CD34+ collection efficiency of hematopoietic progenitor cell collections in sickle cell disease. Transfusion. 2021 Sep;61(9):2775-2781. doi: 10.1111/trf.16551. Epub 2021 Jun 23. PMID 34160085
- [Derived] Boulad F, Shore T, van Besien K, Minniti C, Barbu-Stevanovic M, Fedus SW, Perna F, Greenberg J, Guarneri D, Nandi V, Mauguen A, Yazdanbakhsh K, Sadelain M, Shi PA. Safety and efficacy of plerixafor dose escalation for the mobilization of CD34+ hematopoietic progenitor cells in patients with sickle cell disease: interim results. Haematologica. 2018 May;103(5):770-777. doi: 10.3324/haematol.2017.187047. Epub 2018 Feb 1. PMID 29419425
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/